CLINICAL TRIAL: NCT03352050
Title: Mushroom Effects on Satiety and Gut Health Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1512M81224
Record Dates: First submitted 2017-06-21; First posted 2017-11-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Diet Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ground beef (Active Comparator): ground beef instead of mushrooms
  Interventions: Other: ground beef
- Mushroom (Active Comparator): 2 servings of mushrooms
  Interventions: Dietary Supplement: mushroom

INTERVENTIONS:
Dietary Supplement: mushroom
  Arms: Mushroom
Other: ground beef
  Arms: ground beef

SUMMARY:
The Investigator will compare the effect of mushrooms to ground beef in an intervention study and measure satiety markers and gut health markers

DETAILED DESCRIPTION:
Subjects will consume their habitual diet and the investigators will compare the acute effect of mushroom consumption on satiety and food intake. Additionally, subjects will consume mushrooms for 10 days and the investigators will measure gut health markers, including short chain fatty acids, microbiota, and fecal weight.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Willing to consume mushrooms or ground beef for 10 days

Exclusion Criteria:

* Disease (chronic)
* Smoking,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
satiety | Baseline
  Measure satiety subjectively after consumption of breakfast with mushrooms

SECONDARY OUTCOMES:
Gut health | 10 days
  Measure stool weight and gut microbiota after consumption of mushrooms

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, Principal Investigator — University of Minnesota
Locations (1):
- Department of Food Science and Nutrition, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No